CLINICAL TRIAL: NCT04341935
Title: Effects of DPP4 Inhibition on COVID-19 Patients With Type 2 Diabetes
Brief Title: Effects of DPP4 Inhibition on COVID-19
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Logistical challenges amid COVID-19 pandemic and lack of financial support
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Gianluca Iacobellis, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200384
Record Dates: First submitted 2020-04-06; First posted 2020-04-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Coronavirus Infection; Type 2 Diabetes
Keywords: COVID-19; SARS-Cov 2; DPP4; Type 2 diabetes
MeSH Terms: conditions — Coronavirus Infections; Diabetes Mellitus, Type 2; COVID-19 | interventions — Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DPP4 group (Experimental): Participants in the Dipeptidyl Peptidase 4 (DPP4) group will receive Linagliptin in addition to standard of care insulin regimen as per hospital protocol during hospitalization for up to 14 days
  Interventions: Drug: Linagliptin
- Control group (Active Comparator): Participants in the control group will receive only the standard of care insulin regimen as per hospital protocol during hospitalization for up to 14 days
  Interventions: Drug: Insulin regimen

INTERVENTIONS:
Drug: Linagliptin — 5 mg Linagliptin administered by mouth once daily
  Other Names: Tradjenta
  Arms: DPP4 group
Drug: Insulin regimen — Standard of care insulin regimen as per hospital protocol
  Arms: Control group

SUMMARY:
The purpose of this research is to see if the DPP4 inhibitor linagliptin, an oral medication commonly used to treat type 2 diabetes,can help with diabetes control and reduce the severity of the COVID-19 infection

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus (T2DM) as per American Diabetes Association (ADA) guidelines
* Age ≥ 18
* Confirmed COVID-19
* Mild COVID-19 defined as any of the following: fever, malaise, cough, headache, sore throat, myalgia, nasal congestion, diarrhea
* Moderate COVID-19 is defined as > 2 of the following in non-intubated patients: any symptom of mild disease, radiographic imaging (chest x-ray or lung ultrasound) with bilateral ground glass opacities or bilateral consolidations, SpO2 <90% up to 5L Nasal Cannula (NC)
* No additional signs or symptoms of severe COVID-19.

Exclusion Criteria:

* Type 1 Diabetes Mellitus (T1DM) diabetes, as per ADA guidelines
* History of Diabetic Ketoacidosis (DKA)
* History of acute pancreatitis
* Chronic or Acute Renal Failure with Estimated Glomerular Filtration Rate (eGFR) < 30 ml/min/1.73 m2

Exclusion Criteria:

T1DM diabetes, as per ADA guidelines, History of DKA, History of acute pancreatitis; Chronic or Acute Renal Failure with eGFR < 30 ml/min/1.73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Glucose Llevels | Baseline, up to 2 weeks
  Change in glucose control will be assessed via glucose levels obtained from blood serum samples

SECONDARY OUTCOMES:
Changes in SpO2 levels | Baseline, up to 2 weeks
  changes in SpO2 will be measured with a Pulseimetry, an indirect, non-invasive method
Changes in Interleukin 6 (IL6) | Baseline, up to 2 weeks
  Changes in IL 6 will be assessed from blood serum samples
Changes in chest structures | Baseline, up to 2 weeks
  Changes in Chest radiography (X-ray)

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Iacobellis, MD PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vankadari N, Wilce JA. Emerging WuHan (COVID-19) coronavirus: glycan shield and structure prediction of spike glycoprotein and its interaction with human CD26. Emerg Microbes Infect. 2020 Mar 17;9(1):601-604. doi: 10.1080/22221751.2020.1739565. eCollection 2020. PMID 32178593
- [Result] Iacobellis G. COVID-19 and diabetes: Can DPP4 inhibition play a role? Diabetes Res Clin Pract. 2020 Apr;162:108125. doi: 10.1016/j.diabres.2020.108125. Epub 2020 Mar 26. No abstract available. PMID 32224164